CLINICAL TRIAL: NCT02244151
Title: Evaluation of the Time Interval Between Ovulation Trigger With Triptorelin Acetate and Oocyte Retrieval in IVF Cycles: A Simple Blind, Randomized Controlled Trial.
Brief Title: Evaluation of Time Interval Between Ovulation Trigger With Triptorelin Acetate and Oocyte Retrieval
Acronym: TIMING
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIMING; 2012-005571-14 (EudraCT Number)
Record Dates: First submitted 2014-06-17; First posted 2014-09-18 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2017-08

CONDITIONS: Female Urogenital Diseases
Keywords: ovulation induction,oocyte maturation timing and collection
MeSH Terms: conditions — Female Urogenital Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- DECAPEPTYL® diario (Experimental): Group 1: DECAPEPTYL® diario,OPU 24 hours after GnRHa administration.
  Interventions: Drug: Decapeptyl® diario
- Decapeptyl® diaro (Experimental): Group 2:Decapeptyl® diario OPU 30 hours after GnRHa administration.
  Interventions: Drug: Decapeptyl® diario
- Decapeptyl® diario. (Experimental): Group 3: Decapeptyl® diario, OPU 40 hours after GnRHa administration.
  Interventions: Drug: Decapeptyl® diario
- Decapeptyl® daily (Active Comparator): Group 4: Decapeptyl® daily OPU 36 hrs after GnRH administration
  Interventions: Drug: Decapeptyl® daily

INTERVENTIONS:
Drug: Decapeptyl® diario — Decapeptyl® daily administration (Triptorelin acetate) and follicular puncture at 24, 30, 36 or 40 after administration.
  Other Names: Decapeptyl® daily; GnRHa
  Arms: DECAPEPTYL® diario; Decapeptyl® diario.; Decapeptyl® diaro
Drug: Decapeptyl® daily — Decapeptyl® daily OPU 36 hrs after GnRH administration
  Other Names: Decapeptyl® diario; GnRHa
  Arms: Decapeptyl® daily

SUMMARY:
The aim of this study is to determine what is the best time interval between GnRH agonist (triptorelin acetate) ovulation induction allowing for the higher number of mature oocytes (MII) collected in IVF cycles.

DETAILED DESCRIPTION:
Human chorionic gonadotrophin (hCG) has been the gold standard for ovulation induction for several decades. When GnRH antagonist protocols were introduced, it became possible to trigger final oocyte maturation and ovulation with a single bolus of a GnRH agonist (GnRHa) as an alternative to hCG. The use of GnRHa to trigger final oocyte maturation has potential advantages: the simultaneous induction of a FSH surge, higher numbers of mature oocytes retrieved as compared to hCG and the total elimination of ovarian hyperstimulation syndrome.

From the earliest reports of GnRHa for ovulation triggering, it has been presumed that the timing of the ovum pick-up (OPU) after GnRHa administration should be the same as after hCG triggering (34-36 h). However, differences exist regarding the duration and profile of the GnRHa induced surge of gonadotrophins when compared with that of hCG. Even more, differences in the intra-follicular mechanisms involved in ovulation have been described after GnRHa and hCG trigger.

No previous randomized controlled trials have been reported to evaluate the optimal interval of time between ovulation induction by GnRHa and oocyte collection.

The present study compares the ovarian response and the IVF outcomes after induction by triptorelin 0.2 mg at four different time intervals:

Group 1: OPU 24 hours after GnRHa administration. Group 2: OPU 30 hours after GnRHa administration. Group 3: OPU 40 hours after GnRHa administration. Group 4: control group: OPU 36 hours after GnRHa administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to carry out any procedure associated with the clinical trial.
* Women between 18 and 37 years of age at the time of randomization (both ages included).

Basal serum levels of FSH <10 mIU /ml.

* Serum AMH > 5 to <45 pmol / l.
* Antral follicle count > 6 and < 24.
* Vaginal ultrasound documenting correct visualization of both ovaries and the absence of significant ovarian pathology.
* Short stimulation protocol with GnRH antagonist and conventional dose for ovarian stimulation with 225-300 UI of rhFSH.
* Number of follicles ≥ 16 mm > 5 on the ovulation induction day.

Exclusion Criteria:

* Presence of severe endometriosis (Grade III-IV).
* Absence of one ovary due to previous surgery.
* Presence of significant uterine pathology (submucous myomas, endometrial polyp, malformations..)
* Diagnosis of polycystic ovary syndrome (defined according to the Rotterdam criteria).
* History of previous poor response to conventional ovarian stimulation protocols (< 3 MII oocytes or canceled cycle)
* Severe male factor ( TMS< 1 million).
* Participation in another RCT within the past one year.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2014-09; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes 24 hours post Decapeptyl administration | 24 hours post Decapeptyl administration
  The trial pretends to determine the interval time needed for final oocyte maturation and ovulation after triptorelin administration.
Number of mature oocytes 30 hours post Decapeptyl administration | 30 hours post Decapeptyl administration
  The trial pretends to determine the interval time needed for final oocyte maturation and ovulation after triptorelin administration.
Number of mature oocytes 36 hours post Decapeptyl administration | 36 hours post Decapeptyl administration
  The trial pretends to determine the interval time needed for final oocyte maturation and ovulation after triptorelin administration.
Number of mature oocytes 40 hours post Decapeptyl administration | 40 hours post Decapeptyl administration
  The trial pretends to determine the interval time needed for final oocyte maturation and ovulation after triptorelin administration.

SECONDARY OUTCOMES:
Total number of follicles > 16 mm punctured. | Time 0 (when Decapeptyl administration)
  Total number of follicles > 16 mm punctured.
Total number of oocytes retrieved | 24, 30, 36 and 40 hours post Decapeptyl administration
  Total number of oocytes retrieved
Serum and follicular fluid levels of Amphiregulin (AR) and Epiregulin | 24, 30, 36 and 40 hours post Decapeptyl administration
  Serum and follicular fluid levels of Amphiregulin (AR) and Epiregulin
Serum and follicular fluid hormonal levels (estradiol , LH and progesterone) | Time 0 (when Decapeptyl administration) , 12 hours after Decapeptyl administration , OPU moment and day of embryo transfer
  Serum and follicular fluid hormonal levels (estradiol , LH and progesterone)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Marzal, M.D, Principal Investigator — Grupo de Investigación en Medicina Reproductiva, IIS La Fe, Valencia ; Spain; César Díaz-García, M.D, Study Chair — Unidad de Reproducción Humana, Area de Salud de la Mujer, Hospital Universitaria La Fe, Valencia, Spain. Grupo de Investigación en Medicina Reproductiva, IIS La Fe, Valencia ; Spain; Antonio Pellicer, Professor, Study Director — Unidad de Reproducción Humana, Area de Salud de la Mujer, Hospital Universitaria La Fe, Valencia, Spain. Grupo de Investigación en Medicina Reproductiva, IIS La Fe, Valencia ; Spain.
Locations (1):
- Instituto de Investigacion Sanitaria La Fe, Valencia, Spain